CLINICAL TRIAL: NCT04861129
Title: Bowen Therapy for Chronic Non-specific Low Back Pain: Randomized Controlled Trial
Brief Title: Bowen Therapy for Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: United Christian Hospital (Other)
Responsible Party: Principal Investigator, Andy Shu Kei CHENG, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT_BT_2021
Record Dates: First submitted 2021-04-17; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pain, Back
Keywords: Bowen therapy; Fascia; Low back pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding of participants and outcome assessor will be adopted. Independent assessors who conduct outcome measures are blinded to the group assignments, so allocation concealment and masking can be preserved throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen therapy group (Experimental): The experimental group will receive Bowen therapy according to ISBT Bowen Therapy® (Black & Murray, 2005). It may include sequences 1, 4, 2, hamstrings (movements 1-6) and sacrum sequences in the prone position, and hamstrings sequence (7-18 movements) and 3 in the supine position,. The sequences may also include Bowen movements in the scalenes, trapezius, all erector spinae, sacro-iliac joint ligaments, gluteus maximus and medius, tensor fasciae latae, and gastrocnemius. The application of Bowen sequences is varied between sessions and participants depending on the presenting functional deficit and treatment response.
  Interventions: Procedure: Bowen therapy
- Sham Bowen Therapy group (Sham Comparator): The control group will receive a sham Bowen therapy with the same number of treatment session, treatment time and rest time, that received in the experimental group. However, it consists of gently placing the hands over the areas just enough to maintain contact for the desired time as required by Bowen Therapy, without applying Bowen movement, which is considered the active principle of this technique.
  Interventions: Procedure: Sham Bowen therapy

INTERVENTIONS:
Procedure: Bowen therapy — Intervention is provided weekly for 6 sessions lasting 30-40 mins per treatment session
  Arms: Bowen therapy group
Procedure: Sham Bowen therapy — Sham Intervention is provided weekly for 6 sessions lasting 30-40 mins per treatment session
  Arms: Sham Bowen Therapy group

SUMMARY:
There is emerging evidence that Bowen Therapy may improve musculoskeletal pain. While it can be an effective treatment strategy to enhance pain modulation; studies on the clinical effect are scarce. The aim of this study is to examine the effectiveness of Bowen therapy for people with chronic LBP on measures of pain, function, pain-related self-efficacy, and health related quality of life.

Parallel-group randomized controlled trial (RCT) study will be employed. Pain Catastrophizing Scale (PCS) will be adopted as a screening test upon the randomization. A cutoff of more than 30 points will be used to represents clinically relevant level of catastrophizing.

46 participants with informed consent who meet the eligibility criteria of study are recruited and randomly assigned to one of two groups i.e. Bowen Therapy group and Sham Bowen Conventional Therapy group. Permuted block randomization is applied to control the key confounding variable of catastrophizing which is significantly associated with pain and disability in chronic LBP. Sequentially numbered, opaque, sealed envelopes (SNOSE) is used to ensure the allocation sequence before the group allocation. Double blinding of participants and outcome assessor will be adopted. Measurements are collected at the baseline (Week 0), post-intervention (Week 6) and at a 4-week follow-up (Week 10). The primary outcomes are pain as measured by Percentage of Pain Intensity Difference (PID) and pain relief scale (PRS). The secondary outcomes are measuring the physical functioning, self-efficacy in pain and HRQoL using Owestry Disability Index (ODI), Pain Self-efficacy Questionnaire (PSEQ) and SF-12 (HK) respectively. Intervention is provided weekly for 6 sessions lasting 30-40 minutes per treatment session. The experimental group will receive Bowen therapy according to ISBT Bowen Therapy®. The control group will receive a usual OT therapy with the same number of treatment session, treatment time, including back care advice and functional rehab training.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common condition resulting in socioeconomic burden on health care systems. LBP is defined as pain, muscle tension, or stiffness in the area between the lower posterior margin of the rib cage and the horizontal gluteal fold with or without leg pain. Acute LBP is defined as pain that lasts less than 6 weeks, sub-acute LBP lasts for 6 to 12 weeks, and chronic LBP lasts for longer than 12 weeks. Prevalence study in Hong Kong showed that an estimated 57.1% and 42.1% of the population reported of LBP at least once in their life time and at least once within the past year respectively. In the past decades, several multidisciplinary clinical guidelines were developed in Canada, UK and US for the management of LBP which aimed to promote consistent best practice in patient care. All the guidelines recommended exercise therapy as one the strategy in terms of non-pharmacological, non-invasive management. The National Institute for Health and Care Excellence (NICE) guideline suggested that group exercise programme (biomechanical, aerobic, mind-body or a combination of approaches) should be provided for people with single episode or flare-up of LBP with or without sciatica. Whereas manual therapy could be offered only alongside exercise. Both US and Canadian guidelines advocated similar recommendations. However, none of the guidelines were able to specify which forms of manual therapy is superior for the management of chronic LBP. Bowen therapy is a complementary and alternative medicine involving light touch over the fascial, specific muscles, tendons and connective tissues to improve flow of blood, lymph and energy. It is one of the fascial techniques which aims to release the muscle tension, improve pain and restore function. Bowen therapy was named after Tom Bowen (1916-1982) and also known as Bowen Technique, Bowenwork and Bowtech which are interchangeable in the literature. It promotes connective tissues to slide over each other and improve the afferents responses in response to dysfunction. While Bowen therapy can be an effective treatment strategy to enhance pain modulation; studies on the mechanism of action of Bowen therapy and its clinical effect are scarce.

In most instances, the basic Bowen moves are applied using the fingers and thumbs. It involves taking a slack over skin, applying a gentle non-invasive pressure over muscles, tendon and fascia. Other techniques including fast release, gentle stretching, repetitive squeezing will be used according to the therapist's assessment. Bowen therapy could facilitate tissue hydration and recoiling properties of fascia. It was suggested that Bowen moves in slow release can activate various sensory receptors (e.g. Merkel's Discs, Meissner's corpuscles and Free Nerve Endings) and mechanoreceptors (e.g. Golgi tendon organs, Ruffini endings and Interstitial receptors). For the Bowen moves in fast release, Pacini corpuscles can be activated. The activation of various Golgi tendon organs can lower the sympathetic nervous system (SNS) activity. Furthermore, interstitial receptors stimulated by Bowen moves can also lower SNS and increase vagal tone to achieve the deep relaxing effect and reduction of nerve pressure. It is suggested to adopt different treatment technique of approach to target the dysfunction arising from various types of fascia. The deep fasciae and the epymisium are related to adjustment in coordination, proprioception, balance, myofascial pain, and muscle cramps. According to different anatomical locations and fascial tissue, enough pressure with manual deep friction is required in order to reach the deep fasciae and epymisium. It can explain why some Bowen moves (e.g. Hamstring sequence on biceps femoris) using elbow instead of fingers to exert enough pressure on the soft tissue. Yet in most instances, light massage, which can be achieved in most of the basic Bowen moves, are adequate to address the pain caused by superficial fascia. The Bowen moves also follows a planned sequence of stimulation based on the evidence on myofascial continuity. In Bowen therapy session, two-minute pauses are applied between a set of Bowen moves, that muscle spindles are activated upon the stretch on the muscle fibers. It can be explained by the general pain sensitization of nerve pathways commonly found in people with chronic pain, and so two-minute waiting time allows the body to make appropriate adjustments to re-align and balance, through the mediation at the spinal cord and central nervous system.

Although clinical practice implies that Bowen therapy is a useful technique, particularly in relation to improved pain, joint mobility and functional status; there is still little published research in the literature about the clinical effect of Bowen therapy. Moreover, majority of the studies reviewed lack of control group design and methodological issues, including small sample size, poor sampling method, inadequate information of study sample, and lack of standardized measurement tools. More vigorous and stringent research design is warranted for the future research study.

ELIGIBILITY:
Inclusion Criteria:

* ages between 18 and 65 years
* a diagnosis of low back pain with onset > 12 weeks based on the evaluation by physician
* average pain intensity score of ≥ 3 on NPRS.

Exclusion Criteria:

* they have acute disc prolapse or protusion with neurological sign and symptoms in the past 3-months;
* bacterial spondylitis;
* Rheumatoid arthritis;
* ankylosing spondylitis;
* back pain secondary to bone malignancy
* spinal fracture;
* osteoporotic collapse;
* cauda equina compression
* prior spinal surgery;
* psychiatric disorder (e.g. psychosis / delusion);
* current pregnancy
* previous experience with Bowen therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Percentage of Pain Intensity | Week 6 (compared to Week 0)
  11-point scale by reporting a number from 0 - 10, with "0' representing "no pain" and "10" representing the "most intense pain imaginable". Therefore, the change in pain intensity is expressed as the percentage of pain intensity difference (%PID), which converts the raw score change to a proportional measure i.e. pain intensity difference between the assessments / Pain NRS at baseline assessment. (Score: 0 - 100%)
Change of Percentage of Pain Intensity | Week 10 (compared to Week 0)
  11-point scale by reporting a number from 0 - 10, with "0' representing "no pain" and "10" representing the "most intense pain imaginable". Therefore, the change in pain intensity is expressed as the percentage of pain intensity difference (%PID), which converts the raw score change to a proportional measure i.e. pain intensity difference between the assessments / Pain NRS at baseline assessment. (Score: 0 - 100%)
Pain relief scale | Week 0
  11-point scale with "0" representing "no relief of pain" and "10" representing "completely relieved" to measure the magnitude of change in pain intensity after the treatment. (Score: 0 - 100%)
Pain relief scale | Week 6
  11-point scale with "0" representing "no relief of pain" and "10" representing "completely relieved" to measure the magnitude of change in pain intensity after the treatment. (Score: 0 - 100%)
Pain relief scale | Week 10
  11-point scale with "0" representing "no relief of pain" and "10" representing "completely relieved" to measure the magnitude of change in pain intensity after the treatment. (Score: 0 - 100%)

SECONDARY OUTCOMES:
Owestry Disability Index | Week 0
  Each section has scored from 0 to 5, with 0 representing "no disability" and 5 representing "greatest disability", yielding a total possible score of 50. Finally the score multiplied by two to obtain the index (Score: 0 to 100).
Owestry Disability Index | Week 6
  Each section has scored from 0 to 5, with 0 representing "no disability" and 5 representing "greatest disability", yielding a total possible score of 50. Finally the score multiplied by two to obtain the index (Score: 0 to 100).
Owestry Disability Index | Week 10
  Each section has scored from 0 to 5, with 0 representing "no disability" and 5 representing "greatest disability", yielding a total possible score of 50. Finally the score multiplied by two to obtain the index (Score: 0 to 100).
Chinese version of Pain Self-efficacy Questionnaire | Week 0
  It comprised of 10 items which was rated on a 7-point scale ranging from 0 equals "not at all confident" to 6 equals "completely confident". The total score is calculated by summing up all the items, yielding a maximum possible score of 60. The higher PSEQ score indicated that patients with higher self-efficacy beliefs on performing activities. (Scoring 0 - 60)
Chinese version of Pain Self-efficacy Questionnaire | Week 6
  It comprised of 10 items which was rated on a 7-point scale ranging from 0 equals "not at all confident" to 6 equals "completely confident". The total score is calculated by summing up all the items, yielding a maximum possible score of 60. The higher PSEQ score indicated that patients with higher self-efficacy beliefs on performing activities. (Scoring 0 - 60)
Chinese version of Pain Self-efficacy Questionnaire | Week 10
  It comprised of 10 items which was rated on a 7-point scale ranging from 0 equals "not at all confident" to 6 equals "completely confident". The total score is calculated by summing up all the items, yielding a maximum possible score of 60. The higher PSEQ score indicated that patients with higher self-efficacy beliefs on performing activities. (Scoring 0 - 60)
12-item Chinese (Hong Kong) Short Form Health Survey (version 2) | Week 0
  Higher component summary scores indicate better health and better HRQoL. Range of 0-100 (zero indicating the poorest level of health measured and 100 indicating the highest)
12-item Chinese (Hong Kong) Short Form Health Survey (version 2) | Week 6
  Higher component summary scores indicate better health and better HRQoL. Range of 0-100 (zero indicating the poorest level of health measured and 100 indicating the highest)
12-item Chinese (Hong Kong) Short Form Health Survey (version 2) | Week 10
  Higher component summary scores indicate better health and better HRQoL. Range of 0-100 (zero indicating the poorest level of health measured and 100 indicating the highest)

CONTACTS AND LOCATIONS:
Overall Officials: Andy S.K. Cheng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- United Christian Hospital, Kwun Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: No